CLINICAL TRIAL: NCT00000409
Title: Spine Patient Outcomes Research Trial (SPORT): A Multicenter Randomized Trial for Degenerative Spondylolisthesis (DS) With Spinal Stenosis (SpS) at L4/L5 Level.
Brief Title: Spine Patient Outcomes Research Trial (SPORT): Degenerative Spondylolisthesis With Spinal Stenosis
Acronym: SPORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency); Office of Research on Women's Health (ORWH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01 AR45444 NIAMS-004A; U01AR045444 (NIH)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Spondylolisthesis; Spinal Stenosis; Low Back Pain
Keywords: Intervertebral disc herniation (IDH); Degenerative spondylolisthesis (DS); Spinal stenosis (SpS); Low back pain (LBP); Leg pain; Surgical therapy; Randomized study; Multicenter; MRI; Nonsurgical therapy
MeSH Terms: conditions — Spondylolisthesis; Spinal Stenosis; Low Back Pain; Intervertebral Disc Displacement | interventions — Laminectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery (Active Comparator): Decompressive Laminectomy Fusion-Instrumented Fusion-Non-instrumented
  Interventions: Procedure: Decompressive laminectomy; Other: Non-surgical treatments; Procedure: Fusion--Instrumented; Procedure: Fusion-Non-instrumented
- Non-surgical intervention (Active Comparator): Other. Non-surgical treatments
  Interventions: Other: Non-surgical treatments

INTERVENTIONS:
Procedure: Decompressive laminectomy — Removal of the hypertrophic inferior and superior articular facets will be performed when they are intruding upon the midline and causing both central and lateral recess stenosis
  Arms: Surgery
Other: Non-surgical treatments — Active physical therapy modality, Education/Counseling with home exercise instruction, and an NSAID if tolerated. Any non-operative therapies other than these are accepted and collected as data.
Procedure: Fusion--Instrumented — In addition to decompressive laminectomy, additional bilateral non-instrumented or instrumented, i.e., posterior pedicle fixation, posterolateral fusion with autogenous bone grafting (utilizing iliac crest harvested from between the tables and/or local bone) will be performed between the transverse processes and the lateral portion of the superior facets of the involved levels.
  Arms: Surgery
Procedure: Fusion-Non-instrumented — additional bilateral non-instrumented or instrumented, i.e., posterior pedicle fixation, posterolateral fusion with autogenous bone grafting (utilizing iliac crest harvested from between the tables and/or local bone) will be performed between the transverse processes and the lateral portion of the superior facets of the involved levels.
  Arms: Surgery

SUMMARY:
This study tests the effectiveness of different treatments for the three most commonly diagnosed conditions of the lower backbone (lumbar spine). The purpose is to learn which of two commonly prescribed treatments (surgery and nonsurgical therapy) works better for specific types of low back pain.

In this part of the study, we will treat patients with spinal stenosis (a narrowing of spaces in the backbone that results in pressure on the spinal cord and/or nerve roots) caused by degenerative spondylolisthesis (a condition in which one vertebra, or spinal bone, slips forward on another) with either surgery or nonsurgical methods. This study does not cover the cost of treatment.

DETAILED DESCRIPTION:
Low back pain is considered one of the most widely experienced health problems in the U.S. and the world. It is the second most frequent condition, after the common cold, for which patients see a physician or lose days from work. Estimated costs to those who are severely disabled from low back pain range from $30-70 billion annually. Rates of spinal surgery in the U.S. have increased sharply over time, and researchers have documented 15-fold geographic variation in rates of these surgeries. In many cases, where one lives and who one sees for the condition appear to determine the rates of surgery. Despite these trends, there is little evidence proving the effectiveness of these therapies over nonsurgical management.

This study will use the National Spine Network to conduct a multicenter, randomized, controlled trial for the three most common diagnostic groups for which spine surgery is performed: lumbar intervertebral disc herniation (IDH), spinal stenosis (SpS), and spinal stenosis secondary to degenerative spondylolisthesis (DS). This arm of the trial will deal with patients from the third diagnostic group. The study will compare the most commonly used standard surgical treatments to the most commonly used standard nonsurgical treatments. We will conduct the study at 12 sites throughout the United States.

The primary endpoint of the study will be changes in health-related quality of life as measured by the SF-36 health status questionnaire. Secondary endpoints will include patient satisfaction with treatment, utility for current health in order to estimate quality-adjusted life years (QALYS) as the measure for cost-effectiveness, resource use, and cost.

We will follow patients at 6 weeks and 3, 6, 12, and 24 months to determine their health status, function, satisfaction, and health care use. We anticipate that we will enroll and randomly allocate a total of 300 study participants in this arm of the trial. We will track an additional observational cohort to assess health and resource outcomes. Enrollment in the Observational cohort has been completed as of February 2003.

We will integrate data from the trial and observational cohorts to formally estimate the cost-effectiveness of surgical versus nonsurgical interventions for IDH, SpS, and DS. The results of this trial will provide, for the first time, scientific evidence as to the relative effectiveness of surgical versus nonsurgical treatment for these three most commonly diagnosed lumbar spine conditions.

ELIGIBILITY:
Inclusion Criteria:

* Duration of Symptoms: 12 or more weeks.
* Treatments Tried: Nonsteroidal. anti-inflammatory medical therapy and physical therapy.
* Surgical Screening: Pain in low back, buttocks, or lower extremity that becomes worse with lumbar extension. Must be confirmed by evidence of central or central-lateral compression of the cauda equina by a degenerative lesion of the facet joint, disc, or ligamentum flavum on MRI, computed tomography scans, or myelograms.
* Tests: MRI to confirm diagnosis and level(s).

Exclusion Criteria:

* Previous lumbar spine surgery.
* Not a surgical candidate for any of these reasons: Overall health that makes spinal surgery too life-threatening to be an appropriate alternative, patient has improved dramatically with conservative care, or the patient is unable (for any reason) to undergo surgery within 6 months.
* Possible pregnancy.
* Active malignancy: Patients with a history of any invasive malignancy (except nonmelanoma skin cancer) are ineligible unless they have been treated with curative intent AND have not had any clinical signs or symptoms of the malignancy for at least 5 years.
* Current fracture, infection, and/or deformity (greater than 15 degrees of lumbar scoliosis, using Cobb measure technique) of the spine.
* Age less than 18 years.
* Cauda equina syndrome or progressive neurologic deficit (usually requiring urgent surgery).
* Unavailability for followup (planning to move, no telephone, etc.) or inability to complete data surveys.
* Symptoms less than 12 weeks.
* Patient currently enrolled in any experimental "spine related" study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2000-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Changes in health-related quality of life as measured by the SF-36 health status questionnaire | Baseline, 6 wks, 3 and 6 mos, Annually thereafter

SECONDARY OUTCOMES:
Patient satisfaction with treatment | Baseline, 6 wks, 3 mos, Annually thereafter
utility for current health in order to estimate quality-adjusted life years (QALYS) as the measure for cost effectiveness | Baseline, 1 yr, 4 yr
resource utilization | Baseline, 6 wks, 3 and 6 mos, Annually thereafter
cost | Baseline, 6 wks, 3 and 6 mos, Annually thereafter

CONTACTS AND LOCATIONS:
Overall Officials: James N. Weinstein, DO, MS, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (13):
- United States (13):
  - Kaiser Permanente Spine Care Program, Oakland, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Emory University, The Emory Clinic, Decatur, Georgia
  - Rush-Presbyterian, St. Luke's Medical Center, Chicago, Illinois
  - Maine Spine & Rehabilitation, Scarborough, Maine
  - William Beaumont Hospital, Royal Oak, Michigan
  - Washington University, St Louis, Missouri
  - Nebraska Foundation for Spinal Research, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center - Spine Center, Lebanon, New Hampshire
  - New York University, The Hospital for Joint Diseases, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Rothman Institute at Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Birkmeyer NJ, Weinstein JN, Tosteson AN, Tosteson TD, Skinner JS, Lurie JD, Deyo R, Wennberg JE. Design of the Spine Patient outcomes Research Trial (SPORT). Spine (Phila Pa 1976). 2002 Jun 15;27(12):1361-72. doi: 10.1097/00007632-200206150-00020. PMID 12065987
- [Background] Weinstein JN, Brown PW, Hanscom B, Walsh T, Nelson EC. Designing an ambulatory clinical practice for outcomes improvement: from vision to reality--the Spine Center at Dartmouth-Hitchcock, year one. Qual Manag Health Care. 2000 Winter;8(2):1-20. doi: 10.1097/00019514-200008020-00003. PMID 10787504
- [Background] Fanciullo GJ, Hanscom B, Weinstein JN, Chawarski MC, Jamison RN, Baird JC. Cluster analysis classification of SF-36 profiles for patients with spinal pain. Spine (Phila Pa 1976). 2003 Oct 1;28(19):2276-82. doi: 10.1097/01.BRS.0000084880.33281.EB. PMID 14520044
- [Background] Lurie JD, Birkmeyer NJ, Weinstein JN. Rates of advanced spinal imaging and spine surgery. Spine (Phila Pa 1976). 2003 Mar 15;28(6):616-20. doi: 10.1097/01.BRS.0000049927.37696.DC. PMID 12642771
- [Background] Walsh TL, Hanscom B, Lurie JD, Weinstein JN. Is a condition-specific instrument for patients with low back pain/leg symptoms really necessary? The responsiveness of the Oswestry Disability Index, MODEMS, and the SF-36. Spine (Phila Pa 1976). 2003 Mar 15;28(6):607-15. doi: 10.1097/01.BRS.0000050654.97387.DF. PMID 12642770
- [Result] Weinstein JN, Lurie JD, Tosteson TD, Hanscom B, Tosteson AN, Blood EA, Birkmeyer NJ, Hilibrand AS, Herkowitz H, Cammisa FP, Albert TJ, Emery SE, Lenke LG, Abdu WA, Longley M, Errico TJ, Hu SS. Surgical versus nonsurgical treatment for lumbar degenerative spondylolisthesis. N Engl J Med. 2007 May 31;356(22):2257-70. doi: 10.1056/NEJMoa070302. PMID 17538085
- [Result] Weinstein JN, Lurie JD, Tosteson TD, Zhao W, Blood EA, Tosteson AN, Birkmeyer N, Herkowitz H, Longley M, Lenke L, Emery S, Hu SS. Surgical compared with nonoperative treatment for lumbar degenerative spondylolisthesis. four-year results in the Spine Patient Outcomes Research Trial (SPORT) randomized and observational cohorts. J Bone Joint Surg Am. 2009 Jun;91(6):1295-304. doi: 10.2106/JBJS.H.00913. PMID 19487505
- [Result] Tosteson AN, Tosteson TD, Lurie JD, Abdu W, Herkowitz H, Andersson G, Albert T, Bridwell K, Zhao W, Grove MR, Weinstein MC, Weinstein JN. Comparative effectiveness evidence from the spine patient outcomes research trial: surgical versus nonoperative care for spinal stenosis, degenerative spondylolisthesis, and intervertebral disc herniation. Spine (Phila Pa 1976). 2011 Nov 15;36(24):2061-8. doi: 10.1097/BRS.0b013e318235457b. PMID 22048651
- [Derived] Abdu WA, Lurie JD, Spratt KF, Tosteson AN, Zhao W, Tosteson TD, Herkowitz H, Longely M, Boden SD, Emery S, Weinstein JN. Degenerative spondylolisthesis: does fusion method influence outcome? Four-year results of the spine patient outcomes research trial. Spine (Phila Pa 1976). 2009 Oct 1;34(21):2351-60. doi: 10.1097/BRS.0b013e3181b8a829. PMID 19755935